CLINICAL TRIAL: NCT01576406
Title: A Phase I Study To Evaluate The Effect Of Hepatic Impairment On The Pharmacokinetics And Safety Of Crizotinib In Advanced Cancer Patients
Brief Title: Hepatic Impairment Study For Crizotinib In Advanced Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Basic Science
Other Study IDs: A8081012
Record Dates: First submitted 2012-03-30; First posted 2012-04-12 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-01

CONDITIONS: Advanced Cancer
Keywords: crizotinib; xalkori; PF-02341066; hepatic impairment; pharmacokinetics; advanced cancer
MeSH Terms: interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- A1: normal hepatic function (Experimental)
  Interventions: Drug: crizotinib
- A2: normal hepatic function (Experimental)
  Interventions: Drug: crizotinib
- B: mild hepatic impairment (Experimental)
  Interventions: Drug: crizotinib
- C: moderate hepatic impairment (Experimental)
  Interventions: Drug: crizotinib
- D: severe hepatic impairment (Experimental)
  Interventions: Drug: crizotinib

INTERVENTIONS:
Drug: crizotinib — crizotinib 250 mg twice a day
  Arms: A1: normal hepatic function
Drug: crizotinib — crizotinib 250 mg once a day
  Arms: A2: normal hepatic function
Drug: crizotinib — crizotinib 250 mg twice a day
  Arms: B: mild hepatic impairment
Drug: crizotinib — crizotinib 250 mg once a day
  Arms: C: moderate hepatic impairment
Drug: crizotinib — crizotinib 250 mg once a day
  Arms: D: severe hepatic impairment

SUMMARY:
This study is designed to evaluate the potential effect of hepatic impairment on the pharmacokinetics and safety of crizotinib in advanced cancer patients. Advanced cancer patients with mild, moderate or severe liver dysfunction as well as patients with normal liver function will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid malignancy or lymphoma that is metastatic or unresectable, and for which standard curative or palliative measures do not exist, or are no longer effective. In case of hepatocellular carcinoma, the diagnosis should be based on at least one of the following:

  1. The presence of at least one lesion, measuring ≥ 2 cm, with characteristic arterial enhancement and venous washout in the setting of liver cirrhosis and/or hepatitis B or C infection.
  2. The presence of liver lesion(s) (as defined in a.) with AFP ≥ 400 ng/mL.
  3. Tissue confirmation.
* Biliary obstruction for whom a biliary drain or stent has been placed are eligible, provided that the drain or stent have been in place for at least 10 days prior to the first dose of crizotinib, and the liver function has stabilized as defined by 2 measurements at least 5 days apart that put the patient in the same hepatic dysfunction stratum as defined in Section 3.
* Presence of gliomas and brain metastases only if neurologically stable and treated without ongoing requirement for corticosteroids for at least 2 weeks.
* Any prior systemic therapy (e.g., chemotherapy, molecularly targeted agent, immunotherapy, etc.) or major surgery must have been completed at least 30 days (or as determined by the local requirement, whichever is longer), or at least 5 half lives for drugs with half lives of 6 days or longer prior to initiation of crizotinib treatment. Any prior radiation (except palliative) or minor surgeries/procedures must have been completed at least 2 weeks prior to the initiation of crizotinib treatment. Palliative radiation (≤ 10 fractions) must have been completed 48 hours prior to the initiation of crizotinib treatment. Any acute toxicity must have recovered to Grade ≤1 (except alopecia).
* Eastern Cooperative Oncology Group [ECOG] performance status 0-2.
* Adequate organ function for patients receiving crizotinib therapy as defined by the following criteria:

Bone marrow function

* Absolute neutrophil count (ANC) ≥ 750/uL
* Platelets ≥ 30,000/uL
* Hemoglobin ≥ 8.0 g/dL (≥ 7.0 g/dL for hematologic malignancy) Renal function
* Creatinine ≤ 1.5 x ULN or CrCl > 60 mL/min/1.73 m2 for patients with serum creatinine levels above institutional 1.5 x ULN

  * Male and female patients of childbearing potential must agree to use a highly effective method of contraception throughout the study and for at least 28 days after the last dose of assigned treatment. A patient is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active.

Exclusion Criteria:

* Untreated esophageal varices observed on EGD or imaging study; however, patients with known portal hypertension and evidence of varices on EGD or imaging study who have undergone appropriate therapy as indicated within the last 6 months (if applicable) are eligible for enrollment.
* Uncontrolled ascites that is not stable with medical management (i.e., on diuretics and salt restriction) as defined by requiring therapeutic paracentesis more than once every 4 weeks.
* Episodes of hepatic encephalopathy within the last 4 weeks. Patients with prior episodes of hepatic encephalopathy who are clinically stable on lactulose, neomycin, and/or xifaxan therapy are allowed.
* Prior therapy with crizotinib.
* Spinal cord compression.
* Carcinomatous meningitis or leptomeningeal disease
* Any of the following within the 6 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, or cerebrovascular accident including transient ischemic attack.
* Symptomatic congestive heart failure.
* Ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥ 2, uncontrolled atrial fibrillation of any grade, or an average of triplicate QTc interval >470 msec.
* History of extensive disseminated/bilateral or known presence of interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, and pulmonary fibrosis, but not history of prior radiation pneumonitis.
* Active hemolysis or evidence of biliary sepsis.
* Pregnant females; breastfeeding females; males and females of childbearing potential; males and females of childbearing potential not using highly effective contraception or not agreeing to continue highly effective contraception for at least 28 days after last dose of investigational product; males and females of childbearing potential not using two (2) methods of highly effective contraception or not agreeing to continue two (2) methods of highly effective contraception for at least 28 days after last dose of investigational product.
* Use of drugs or foods that are known strong CYP3A4 inhibitors, including but not limited to atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, troleandomycin, voriconazole, and grapefruit or grapefruit juice.
* Use of drugs that are known strong CYP3A4 inducers, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, and St. John's wort.
* Use of drugs that are CYP3A4 substrates with narrow therapeutic indices, including but not limited to dihydroergotamine, ergotamine, and pimozide.
* Other severe acute or chronic medical (may include severe gastrointestinal conditions such as chronic diarrhea or ulcer disease) or psychiatric conditions, or laboratory abnormalities that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of the study results and, in the judgment of the investigator, would make the patient inappropriate for study entry.
* Patients who had prior major gastrointestinal surgery removing part of gastrointestinal tract and/or gall bladder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (20):
  - Keck Hospital of USC, Los Angeles, California
  - LAC&USC Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center / Investigational Drug Services, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Anschutz Cancer Pavilion, Room 2224, c/o Melinda Friesleben, Pharm D, Aurora, Colorado
  - University of Colorado Denver - Clinical Translational Research Center, Aurora, Colorado
  - University of Colorado Denver, Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado Denver, Anschutz Inpatient Pavillion, Aurora, Colorado
  - Emory University Hospital Midtown Laboratory, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Investigational Drug Service: The Emory Clinic Bldg A, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - University Hospital East, Columbus, Ohio
  - Investigational Drug Services, Columbus, Ohio
  - James Cancer Hospital, Columbus, Ohio
  - The Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Martha Morehouse Medical Plaza, Columbus, Ohio
  - Cancer Therapy & Research Center at UTHSCSA, San Antonio, Texas
  - Medical Arts and Research Center-MARC, San Antonio, Texas

REFERENCES:
- [Derived] El-Khoueiry AB, Sarantopoulos J, O'Bryant CL, Ciombor KK, Xu H, O'Gorman M, Chakrabarti J, Usari T, El-Rayes BF. Evaluation of hepatic impairment on pharmacokinetics and safety of crizotinib in patients with advanced cancer. Cancer Chemother Pharmacol. 2018 Apr;81(4):659-670. doi: 10.1007/s00280-018-3517-8. Epub 2018 Feb 21. PMID 29468455
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081012&StudyName=Hepatic%20Impairment%20Study%20For%20Crizotinib%20In%20Advanced%20Cancer%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Hepatic Function: Crizotinib 250 mg Twice Daily: Participants with normal hepatic function received Crizotinib 250 milligram (mg) capsules, orally, twice daily continuously in 28-day cycles. Treatment was continued until disease progression, unacceptable toxicity or withdrawal of consent occurred. Normal hepatic function was defined as total bilirubin and aspartate aminotransferase (AST) levels less than or equal to (<=) the upper limit of normal (ULN).
- Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily: Participants with normal hepatic function received Crizotinib 200 mg capsules, orally, twice daily continuously in 28-day cycles and dose could be increased to 250 mg twice daily after completion of pharmacokinetic (PK) assessment on Cycle 2 Day 1 based on their tolerability. Treatment was continued until disease progression, unacceptable toxicity or withdrawal of consent occurred. Normal hepatic function was defined as total bilirubin and AST levels <=ULN.
- Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily: Participants with mild hepatic impairment received Crizotinib 250 mg capsules, orally, twice daily continuously in 28-day cycles. Treatment was continued until disease progression, unacceptable toxicity or withdrawal of consent occurred. Mild hepatic impairment was defined as total bilirubin level <=ULN and AST levels greater than (>) ULN or total bilirubin level > 1.0 to 1.5*ULN.
- Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily: Participants with moderate hepatic impairment received Crizotinib 250 mg capsules, orally, once daily continuously in 28-day cycles. Treatment was continued until disease progression, unacceptable toxicity or withdrawal of consent occurred. Moderate hepatic impairment was defined as total bilirubin level >1.5 to 3*ULN
- Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily: Participants with moderate hepatic impairment received Crizotinib 200 mg capsules, orally, twice daily continuously in 28-day cycles. Treatment was continued until disease progression, unacceptable toxicity or withdrawal of consent occurred. Moderate hepatic impairment was defined as total bilirubin level >1.5 to 3*ULN
- Severe Hepatic Impairment Crizotinib 250 mg Once Daily: Participants with severe hepatic impairment received Crizotinib 250 mg capsules, orally, once daily continuously in 28-day cycles. Treatment was continued until disease progression, unacceptable toxicity or withdrawal of consent occurred. Severe hepatic Impairment was defined as total bilirubin level >3*ULN.
Period: Overall Study
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Started | 11 | 15 | 20 | 10 | 16 | 16
Completed | 5 | 7 | 4 | 1 | 8 | 4
Not Completed | 6 | 8 | 16 | 9 | 8 | 12
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 3 | 4 | 8 | 5 | 7 | 9
Not completed — Non-clinical trial supply of Crizotinib | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal the consent | 2 | 2 | 5 | 1 | 1 | 3
Not completed — Other | 0 | 0 | 2 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all enrolled participants who received at least 1 dose of Crizotinib on Cycle 1, Day 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily | Total
Number analyzed (Participants) | 11 | 15 | 20 | 10 | 16 | 16 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (15.64) | 62.9 (10.35) | 61.2 (10.14) | 59.2 (8.85) | 60.3 (7.87) | 59.0 (6.04) | 60.3 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 7 | 2 | 6 | 6 | 31
  Male | 7 | 9 | 13 | 8 | 10 | 10 | 57

OUTCOME MEASURES:

1. Primary Outcome: Area Under Plasma Concentration Time Curve From Time Zero to End of Dosing Interval (AUCtau) of Crizotinib: Cycle 2 Day 1
Description: Area under the plasma concentration-time curve from time zero to the quantifiable concentration at the end of dosing interval (tau hours post-dose, where tau was 12 hours for twice daily dosing and 24 hours for once daily dosing) of Cycle 2 Day 1.
Time Frame: Cycle 2 Day 1- Twice daily dosing: pre-dose and 1, 2, 4, 6, 8, 12 hours post-dose; Once daily dosing: pre-dose and 1, 2, 4, 6, 8, 24 hours post-dose
Population: PK evaluable set:Cycle 2 Day 1(C2D1)full PK collected;no dose change;atleast 14 days of constant dosing before C2D1 or>80% of Crizotinib during 14 days prior to C2D1;not vomited Crizotinib on same day of PK collection on C2D1;no prior major GI surgery;11 days of constant dosing instead of 14 days before C2D1 but met all other PK evaluable criteria.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
nanogram*hour per milliliter (ng*hr/mL) | 3552 (48) | 2712 (66) | 3238 (73) | 2305 (83) | 4057 (58) | 4596 (63)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Crizotinib: Cycle 2 Day 1
Time Frame: as for outcome 1
Population: PK evaluable set: C2D1 full PK collected;no dose change;atleast 14 days of constant dosing before C2D1 or>80% of Crizotinib during 14 days prior to C2D1;not vomited Crizotinib on same day of PK collection on C2D1;no prior major GI surgery;11 days of constant dosing instead of 14 days before C2D1 but met all other PK evaluable criteria.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
nanogram per milliliter (ng/mL) | 375.1 (50) | 283.9 (65) | 342.1 (68) | 152.9 (58) | 408.3 (56) | 272.4 (29)
Statistical Analysis 1: Comparison: Normal Hepatic Function: Crizotinib 250 mg Twice Daily vs Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily; Confidence interval (CI): Geometric mean ratio and 90 percent (%) CI were derived from analysis of variance (ANOVA) model; Test type: Superiority; Geometric mean ratio = 91.20, 90% CI 2-sided [57.47 to 144.72]
Statistical Analysis 2: Comparison: Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily vs Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily; CI: Geometric mean ratio and 90% CI were derived from ANOVA model; Test type: Superiority; Geometric mean ratio = 143.82, 90% CI 2-sided [89.11 to 232.12]
Statistical Analysis 3: Comparison: Normal Hepatic Function: Crizotinib 250 mg Twice Daily vs Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily; CI: Geometric mean ratio and 90% CI were derived from ANOVA model; Test type: Superiority; Geometric mean ratio = 108.87, 90% CI 2-sided [70.13 to 168.99]
Statistical Analysis 4: Comparison: Normal Hepatic Function: Crizotinib 250 mg Twice Daily vs Severe Hepatic Impairment Crizotinib 250 mg Once Daily; CI: Geometric mean ratio and 90% CI were derived from ANOVA model; Test type: Superiority; Geometric mean ratio = 72.63, 90% CI 2-sided [49.07 to 107.50]

3. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Quantifiable Plasma Concentration (AUClast) of Crizotinib: Cycle 1 Day 1
Time Frame: Cycle 1 Day 1- Twice daily dosing: pre-dose and 1, 2, 4, 6, 8, 12 hours post-dose; Once daily dosing: pre-dose and 1, 2, 4, 6, 8, 24 hours post-dose
Population: PK evaluable set. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 9 | 7 | 8 | 6
ng*hr/mL | 732.3 (84) | 520.8 (49) | 557.5 (78) | 610.4 (128) | 684.9 (89) | 856.7 (57)

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Crizotinib: Cycle 1 Day 1
Time Frame: as for outcome 3
Population: PK evaluable set. Here, 'N' signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 9 | 7 | 8 | 6
ng/mL | 101.9 (92) | 84.52 (67) | 102.3 (66) | 57.74 (112) | 99.59 (88) | 90.69 (63)

5. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Crizotinib: Cycle 1 Day 1
Time Frame: as for outcome 3
Population: PK evaluable set. Here, 'N' signifies those participants who were evaluable for this measure.
Measure: Median (Full Range); unit: hour
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 9 | 7 | 8 | 6
hour | 4.00 [1.00 to 6.00] | 4.00 [1.00 to 6.00] | 4.00 [1.92 to 10.9] | 2.02 [1.00 to 4.05] | 4.00 [1.00 to 8.00] | 3.00 [1.00 to 6.00]

6. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of Crizotinib: Cycle 2 Day 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
ng/mL | 238.6 (52) | 170.9 (75) | 179.1 (101) | 47.44 (376) | 287.0 (58) | 135.5 (102)

7. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Quantifiable Plasma Concentration (AUClast) of Crizotinib: Cycle 2 Day 1
Time Frame: as for outcome 1
Population: Data for this outcome measure was not estimated, since few secondary PK parameters listed in the protocol and/or SAP were not estimated, due to change in planned analysis. However, it did not affect the interpretation of the final PK data.
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Plasma Accumulation Ratio (Rac) of Crizotinib
Description: Rac was defined as the ratio of AUCtau of Cycle 2 Day 1 to AUCtau of Cycle 1 Day 1, where AUCtau was area under the plasma concentration-time curve from time zero to the quantifiable concentration at the end of dosing interval (tau hours post-dose, where tau was 12 hours for twice daily dosing and 24 hours for once daily dosing).
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1- Twice daily dosing: pre-dose and 1, 2, 4, 6, 8, 12 hours post-dose; Once daily dosing: pre-dose and 1, 2, 4, 6, 8, 24 hours post-dose
Population: as for outcome 7
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Apparent Oral Clearance (CL/F) of Crizotinib: Cycle 2 Day 1
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent oral clearance was obtained by dividing study drug dose with AUCtau, where AUCtau was area under the plasma concentration-time curve from time zero to the quantifiable concentration at the end of dosing interval (tau hours post-dose, where tau was 12 hours for twice daily dosing and 24 hours for once daily dosing) of Cycle 2 Day 1.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
Liter/hour | 70.39 (48) | 73.79 (66) | 77.21 (73) | 108.5 (83) | 49.26 (58) | 54.36 (63)

10. Secondary Outcome: Fraction of Unbound Crizotinib in Plasma: Cycle 2 Day 1
Description: Fraction of unbound Crizotinib concentration in plasma was defined as the ratio of unbound Crizotinib concentration to the total Crizotinib concentration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
ratio | 0.03624 (26) | 0.03066 (27) | 0.04315 (31) | 0.05406 (20) | 0.04152 (34) | 0.03523 (46)

11. Secondary Outcome: Unbound Area Under the Plasma Concentration Time Curve From Time Zero to the Last Quantifiable Plasma Concentration (AUClast) of Crizotinib: Cycle 2 Day 1
Description: Unbound area under the plasma concentration-time curve from time zero to the last quantifiable plasma concentration post-dose of Cycle 2 day 1.
Time Frame: as for outcome 1
Population: as for outcome 7
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Unbound Area Under Plasma Concentration-Time Curve From Time Zero to End of Dosing Interval (AUCtau) of Crizotinib: Cycle 2 Day 1
Description: Unbound area under the plasma concentration-time curve from time zero to the quantifiable concentration at the end of dosing interval (tau hours post-dose, where tau was 12 hours for twice daily dosing and 24 hours for once daily dosing) of Cycle 2 Day 1.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
ng*hr/mL | 128.7 (38) | 83.08 (73) | 139.7 (94) | 124.6 (85) | 168.6 (59) | 161.9 (48)

13. Secondary Outcome: Unbound Maximum Observed Plasma Concentration (Cmax) of Crizotinib: Cycle 2 Day 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
ng/mL | 13.59 (41) | 8.703 (74) | 14.77 (93) | 8.271 (62) | 16.96 (56) | 9.608 (34)

14. Secondary Outcome: Area Under Plasma Concentration Time Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06260182: Cycle 2 Day 1
Description: Area under the plasma concentration-time curve from time zero to the quantifiable concentration at the end of dosing interval (tau hours postdose, where tau was 12 hours for twice daily dosing and 24 hours for once daily dosing) of Cycle 2 Day 1. AUCtau of PF-06260182, (a metabolite of Crizotinib) is reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
ng*hr/mL | 1087 (43) | 717.4 (81) | 480.3 (168) | 200.0 (48) | 391.8 (118) | 434.0 (96)

15. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Plasma Concentration (AUClast) of PF-06260182: Cycle 1 Day 1
Description: AUClast of PF-06260182, (a metabolite of Crizotinib) is reported in this outcome measure.
Time Frame: as for outcome 3
Population: PK evaluable set. Here, 'N' signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 9 | 7 | 8 | 6
ng*hr/mL | 272.4 (80) | 166.5 (31) | 90.71 (153) | 64.90 (103) | 53.36 (139) | 59.61 (81)

16. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-06260182: Cycle 1 Day 1
Description: Cmax of PF-06260182, (a metabolite of Crizotinib) is reported in this outcome measure.
Time Frame: as for outcome 3
Population: PK evaluable set. Here, 'N' signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 9 | 7 | 8 | 6
ng/mL | 35.48 (86) | 24.12 (33) | 13.54 (153) | 4.869 (95) | 6.995 (152) | 4.088 (88)

17. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-06260182: Cycle 2 Day 1
Description: Cmax of PF-06260182, (a metabolite of Crizotinib) is reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
ng/mL | 108.5 (43) | 73.47 (76) | 50.34 (164) | 12.43 (55) | 39.32 (120) | 25.15 (110)

18. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06260182: Cycle 1 Day 1
Description: Tmax of PF-06260182, (a metabolite of Crizotinib) is reported in this outcome measure.
Time Frame: as for outcome 3
Population: PK evaluable set. Here, 'N' signifies those participants who were evaluable for this measure.
Measure: Median (Full Range); unit: hour
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 9 | 7 | 8 | 6
hour | 6.04 [4.00 to 8.00] | 4.00 [2.00 to 8.00] | 4.00 [4.00 to 10.9] | 6.08 [5.93 to 8.00] | 8.00 [4.00 to 12.00] | 7.00 [4.00 to 8.00]

19. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06260182: Cycle 2 Day 1
Description: Tmax of PF-06260182, (a metabolite of Crizotinib) is reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
hour | 6.00 [0.983 to 10.0] | 4.03 [1.00 to 7.45] | 4.00 [0 to 10.8] | 6.00 [4.05 to 7.30] | 0 [0 to 6.00] | 6.69 [0 to 8.00]

20. Secondary Outcome: Metabolite Ratio for Area Under Plasma Concentration Time Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06260182: Cycle 2 Day 1
Description: Metabolite ratio for AUCtau was defined as the ratio of AUCtau of metabolite (PF-06260182) to AUCtau of parent drug (Crizotinib), where AUCtau was the area under the plasma concentration-time curve from time zero to the quantifiable concentration at the end of dosing interval (tau was 12 hours for twice daily dosing and 24 hours for once daily dosing) of Cycle 2 Day 1.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
ratio | 0.2968 (17) | 0.2569 (31) | 0.1439 (74) | 0.08402 (65) | 0.09360 (47) | 0.09162 (47)

21. Secondary Outcome: Metabolite Ratio for Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Quantifiable Plasma Concentration (AUClast) of PF-06260182: Cycle 1 Day 1
Description: Metabolite ratio for AUClast was defined as the ratio of AUClast of metabolite (PF-06260182) to AUClast of parent drug (Crizotinib), where AUClast was area under the plasma concentration-time curve from time zero to the last quantifiable plasma concentration post-dose of Cycle 1 Day 1.
Time Frame: as for outcome 3
Population: PK evaluable set. Here, 'N' signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 9 | 7 | 8 | 6
ratio | 0.3608 (18) | 0.3104 (30) | 0.1577 (60) | 0.1032 (72) | 0.07566 (42) | 0.06753 (21)

22. Secondary Outcome: Metabolite Ratio for Maximum Observed Plasma Concentration (Cmax) of PF-06260182: Cycle 1 Day 1
Description: Metabolite ratio for Cmax was defined as the ratio of Cmax of metabolite (PF-06260182) to Cmax of parent drug (Crizotinib), where Cmax was maximum observed plasma concentration post-dose of Cycle 1 Day 1.
Time Frame: as for outcome 3
Population: PK evaluable set. Here, 'N' signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 9 | 7 | 8 | 6
ratio | 0.3378 (25) | 0.2769 (41) | 0.1284 (70) | 0.08178 (66) | 0.06809 (47) | 0.04373 (42)

23. Secondary Outcome: Metabolite Ratio for Maximum Observed Plasma Concentration (Cmax) of PF-06260182: Cycle 2 Day 1
Description: Metabolite ratio for Cmax was defined as the ratio of Cmax of metabolite (PF-06260182) to Cmax of parent drug (Crizotinib), where Cmax was maximum observed plasma concentration post-dose of Cycle 2 Day 1.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
ratio | 0.2804 (19) | 0.2511 (31) | 0.1428 (73) | 0.07881 (58) | 0.09337 (49) | 0.08954 (90)

24. Secondary Outcome: Fraction of Unbound PF-06260182 in Plasma: Cycle 2 Day 1
Description: Fraction of unbound PF-06260182 (a metabolite of Crizotinib) in plasma was defined as the ratio of unbound PF-06260182 concentration in plasma to the total PF-06260182 concentration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
ratio | 0.03797 (11) | 0.03822 (16) | 0.04857 (16) | 0.05788 (22) | 0.05031 (10) | 0.05177 (13)

25. Secondary Outcome: Unbound Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Plasma Concentration (AUClast) of PF-06260182: Cycle 2 Day 1
Description: Unbound AUClast of PF-06260182 (a metabolite of Crizotinib) is reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 7
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Unbound Area Under Plasma Concentration Time Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06260182: Cycle 2 Day 1
Description: Unbound area under the plasma concentration-time curve from time zero to the quantifiable concentration at the end of dosing interval (tau hours post-dose, where tau was 12 hours for twice daily dosing and 24 hours for once daily dosing) of Cycle 2 Day 1. Unbound AUCtau of PF-06260182, (a metabolite of Crizotinib) is reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
ng*hr/mL | 41.26 (36) | 27.40 (99) | 23.35 (181) | 11.56 (49) | 19.71 (119) | 22.49 (79)

27. Secondary Outcome: Unbound Maximum Observed Plasma Concentration (Cmax) of PF-06260182: Cycle 2 Day 1
Description: Unbound Cmax of PF-06260182, (a metabolite of Crizotinib) is reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
ng/mL | 4.119 (36) | 2.806 (94) | 2.445 (178) | 0.7194 (50) | 1.977 (122) | 1.301 (93)

28. Other Pre Specified Outcome: Area Under the Plasma Concentration Time Curve as Daily Exposure (AUCdaily) of Crizotinib: Cycle 2 Day 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
ng*hr/mL | 7107 (48) | 5422 (66) | 6476 (73) | 2305 (83) | 8108 (58) | 4596 (63)
Statistical Analysis 1: Comparison: Normal Hepatic Function: Crizotinib 250 mg Twice Daily vs Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily; CI: Geometric mean ratio and 90% CI were derived from ANOVA model; Test type: Superiority; Percentage of ratio of geometric mean = 91.12, 90% CI 2-sided [56.56 to 146.79]
Statistical Analysis 2: Comparison: Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily vs Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily; CI: Geometric mean ratio and 90% CI were derived from ANOVA model; Test type: Superiority; Percentage of ratio of geometric mean = 149.54, 90% CI 2-sided [91.85 to 243.46]
Statistical Analysis 3: Comparison: Normal Hepatic Function: Crizotinib 250 mg Twice Daily vs Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily; CI: Geometric mean ratio and 90% CI were derived from ANOVA model; Test type: Superiority; Percentage of ratio of geometric mean = 114.08, 90% CI 2-sided [73.57 to 176.89]
Statistical Analysis 4: Comparison: Normal Hepatic Function: Crizotinib 250 mg Twice Daily vs Severe Hepatic Impairment Crizotinib 250 mg Once Daily; CI: Geometric mean ratio and 90% CI were derived from ANOVA model; Test type: Superiority; Percentage of ratio of geometric mean = 64.67, 90% CI 2-sided [39.50 to 105.89]

29. Other Pre Specified Outcome: Unbound Area Under the Plasma Concentration Time Curve as Daily Exposure (AUCdaily) of Crizotinib: Cycle 2 Day 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
ng*hr/mL | 257.7 (38) | 166.1 (73) | 279.4 (95) | 124.6 (85) | 337.0 (59) | 161.9 (48)
Statistical Analysis 1: Comparison: Normal Hepatic Function: Crizotinib 250 mg Twice Daily vs Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily; CI: Geometric mean ratio and 90% CI were derived from ANOVA model; Test type: Superiority; Percentage of ratio of geometric mean = 108.43, 90% CI 2-sided [63.47 to 185.26]
Statistical Analysis 2: Comparison: Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily vs Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily; CI: Geometric mean ratio and 90% CI were derived from ANOVA model; Test type: Superiority; Percentage of ratio of geometric mean = 202.89, 90% CI 2-sided [120.96 to 340.30]
Statistical Analysis 3: Comparison: Normal Hepatic Function: Crizotinib 250 mg Twice Daily vs Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily; CI: Geometric mean ratio and 90% CI were derived from ANOVA model; Test type: Superiority; Percentage of ratio of geometric mean = 130.78, 90% CI 2-sided [86.61 to 197.47]
Statistical Analysis 4: Comparison: Normal Hepatic Function: Crizotinib 250 mg Twice Daily vs Severe Hepatic Impairment Crizotinib 250 mg Once Daily; CI: Geometric mean ratio and 90% CI were derived from ANOVA model; Test type: Superiority; Percentage of ratio of geometric mean = 62.82, 90% CI 2-sided [42.54 to 92.78]

30. Other Pre Specified Outcome: Area Under the Plasma Concentration Time Curve as Daily Exposure (AUCdaily) of PF-06260182: Cycle 2 Day 1
Description: AUCdaily of PF-06260182, (a metabolite of Crizotinib) is reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
ng*hr/mL | 2173 (43) | 1435 (81) | 961.2 (168) | 200.0 (48) | 784.0 (117) | 434.0 (96)

31. Other Pre Specified Outcome: Unbound Area Under the Plasma Concentration Time Curve as Daily Exposure (AUCdaily) of PF-06260182: Cycle 2 Day 1
Description: Unbound AUCdaily of PF-06260182, (a metabolite of Crizotinib) is reported in this outcome measure, where AUCdaily was area under the plasma concentration time curve as daily exposure post-dose.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 8 | 9 | 10 | 7 | 8 | 6
ng*hr/mL | 82.56 (36) | 54.85 (99) | 46.66 (181) | 11.56 (49) | 39.41 (119) | 22.49 (79)

32. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 4 years that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: From initiation of treatment up to follow-up period (up to 4 years)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 11 | 15 | 20 | 10 | 16 | 16
participants
  AEs | 11 | 15 | 20 | 9 | 16 | 16
  SAEs | 7 | 8 | 13 | 6 | 14 | 14

33. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events, by National Cancer Institute (NCI) Common Terminology Criteria (CTC) for AEs (CTCAE) (Version 4.0) Grade
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE was assessed according to severity grading based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events [CTCAE] Version 4.0. Grade 1 =mild; Grade 2 =moderate; Grade 3 =severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated; Grade 4 =life-threatening or disabling, urgent intervention indicated; Grade 5 =death. Treatment-emergent events were events between first dose of study drug and up to 4 years that were absent before treatment that worsened relative to pretreatment state. If the same participant in a given treatment had more than 1 adverse event, only the maximum CTCAE was reported.
Time Frame: From initiation of treatment up to follow-up period (up to 4 years)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 11 | 15 | 20 | 10 | 16 | 16
participants
  Grade 1 AEs | 1 | 2 | 2 | 0 | 0 | 0
  Grade 2 AEs | 2 | 6 | 5 | 1 | 0 | 1
  Grade 3 AEs | 6 | 3 | 5 | 2 | 9 | 8
  Grade 4 AEs | 0 | 1 | 2 | 1 | 2 | 0
  Grade 5 AEs | 2 | 3 | 6 | 5 | 5 | 7

34. Other Pre Specified Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both serious and non-serious adverse events.
Time Frame: From initiation of treatment up to follow-up period (up to 4 years)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 11 | 15 | 20 | 10 | 16 | 16
participants
  AE | 9 | 14 | 15 | 6 | 11 | 11
  SAE | 0 | 3 | 0 | 0 | 0 | 0

35. Other Pre Specified Outcome: Number of Participants With Laboratory Test Abnormalities: NCI CTCAE (Version 4.0) Grade 1 to 4 Hematological Test Abnormalities
Description: Anemia(grade[g]1:Less than[<] Lower limit of normal[LLN] to 10gram per[/] deciliter[g/dL],g2:<10 to 8g/dL,g3:<8g/dL,g4:lifethreatening);platelet (g1:<LLN to 75*10^3/millimeter[mm]^3,g2:<75*10^3/mm^3 to 50*10^3/mm^3,g3:<50*10^3/mm^3 to 25*10^3/mm^3,g4:<25*10^3/mm^3);lymphopenia(g1:<LLN to 8*10^2/mm^3,g2:<8*10^2 to 5*10^2/mm^3,g3:<5*10^2 to 2*10^2/mm^3,g4:<2*10^2/mm^3);neutrophil (Absolute)(g1:<LLN to 15*10^2/mm^3,g2:<15*10^2 to 10*10^2/mm^3,g3:<10*10^2 to 5*10^2/mm^3,g4:<5*10^2/mm^3);white blood cell count(g1:<LLN to 3*10^3/mm^3,g2:<3*10^3 to 2*10^3/mm^3,g3:<2*10^3 to 1*10^3/mm^3,g4:<1*10^3/mm^3);hemoglobin(g1:increase in hemoglobin level>0 to 2 g/dL above ULN or above baseline if baseline is above ULN,g2:increase in hemoglobin level>2 to 4g/dL above ULN or above baseline if baseline is above ULN,g3:increase in hemoglobin level>4 g/dL above ULN or above baseline if baseline is above ULN). Only categories with atleast 1 participant with abnormality are reported in this outcome measure.
Time Frame: Baseline up to end of treatment (up to 728 days)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 11 | 15 | 20 | 10 | 16 | 16
participants
  Anemia: Grade 1 | 4 | 7 | 9 | 9 | 7 | 8
  Anemia: Grade 2 | 4 | 7 | 4 | 1 | 5 | 5
  Anemia: Grade 3 | 1 | 1 | 3 | 0 | 1 | 1
  Hemoglobin Increased: Grade 1 | 0 | 0 | 1 | 0 | 0 | 0
  Lymphopenia: Grade 1 | 2 | 2 | 5 | 2 | 0 | 1
  Lymphopenia: Grade 2 | 3 | 7 | 4 | 6 | 9 | 7
  Lymphopenia: Grade 3 | 1 | 1 | 3 | 2 | 2 | 4
  Lymphopenia: Grade 4 | 0 | 0 | 0 | 0 | 2 | 0
  Neutrophils (Absolute): Grade 1 | 0 | 0 | 1 | 2 | 1 | 2
  Neutrophils (Absolute): Grade 2 | 3 | 1 | 2 | 0 | 3 | 0
  Neutrophils (Absolute): Grade 3 | 0 | 0 | 1 | 0 | 1 | 3
  Platelets: Grade 1 | 0 | 2 | 4 | 2 | 8 | 3
  Platelets: Grade 2 | 0 | 0 | 1 | 0 | 2 | 2
  Platelets: Grade 3 | 0 | 0 | 2 | 3 | 2 | 5
  White Blood Cells: Grade 1 | 2 | 3 | 4 | 2 | 2 | 1
  White Blood Cells: Grade 2 | 1 | 1 | 3 | 2 | 3 | 3
  White Blood Cells: Grade 3 | 0 | 0 | 0 | 0 | 1 | 3

36. Other Pre Specified Outcome: Number of Participants With Laboratory Test Abnormalities: NCI CTCAE (Version 4.0) Grade 1 to 4 Chemistry Test Abnormalities
Description: ALT/AST(grade[g]1:>ULN-3*ULN,g2:>3-5*ULN,g3:>5-20*ULN,g4:>20*ULN);AP(g1:>ULN-2.5*ULN,g2:>2.5-5*ULN,g3:>5-20*ULN,g4:>20*ULN);CR(g1:>ULN-1.5*ULN,g2:>1.5-3*ULN,g3:>3-6*ULN,g4:>6*ULN);hyperglycemia(g1:>ULN-160mg/dL,g2:>160-250mg/dL,g3:>250-500mg/dL,g4:>500mg/dL);bilirubin(total)(g1:>ULN-1.5*ULN,g2:>1.5-3*ULN,g3:>3-10*ULN,g4:>10*ULN);hypoglycemia(g1:<LLN-55mg/dL,g2:<55-40mg/dL,g3:<40-30mg/dL,g4:<30mg/dL);hyperkalemia(g1:>ULN-5.5mmol/L,g2:>5.5-6mmol/L,g3:>6-7mmol/L,g4:>7mmol/L);hypokalemia(g1:<LLN-3mmol/L,g2:<LLN-3mmol/L,g3:<3-2.5mmol/L,g4:<2.5mmol/L);hypermagnesemia(g1:>ULN-3mg/dL,g3:>3-8mg/dL,g4:>8mg/dL);hypocalcemia(g1:<LLN-8mg/dL,g2:<8-7mg/dL,g3:<7-6mg/dL,g4:<6mg/dL);hypomagnesemia(g1:<LLN-1.2mg/dL,g2:<1.2-0.9mg/dL,g3:<0.9-0.7mg/dL,g4:<0.7mg/dL);hyponatremia(g1:<LLN-130mmol/L,g3:<130-120mmol/L,g4:<120mmol/L);hypoalbuminemia(g1:<LLN-3g/dL,g2:<3-2g/dL,g3:<2g/dL,g4:lifethreatening);hypophosphatemia(g1:<LLN-2.5mg/dL,g2:<2.5-2mg/dL,g3:<2-1mg/dL,g4:<1mg/dL).Participant>=1abnormality given.
Time Frame: Baseline up to end of treatment (up to 728 days)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 11 | 15 | 20 | 10 | 16 | 16
participants
  Alanine aminotransferase (ALT): Grade 1 | 8 | 3 | 12 | 6 | 12 | 9
  ALT: Grade 2 | 0 | 0 | 5 | 2 | 3 | 5
  ALT: Grade 3 | 0 | 0 | 0 | 1 | 1 | 0
  Alkaline phosphatase(AP): Grade 1 | 4 | 7 | 8 | 4 | 7 | 5
  Alkaline phosphatase: Grade 2 | 2 | 1 | 5 | 3 | 4 | 4
  Alkaline phosphatase: Grade 3 | 0 | 1 | 3 | 3 | 4 | 6
  AST:Grade 1 | 6 | 7 | 8 | 5 | 4 | 4
  AST: Grade 2 | 1 | 0 | 7 | 0 | 7 | 3
  AST: Grade 3 | 0 | 1 | 3 | 5 | 5 | 7
  AST: Grade 4 | 0 | 0 | 0 | 0 | 0 | 2
  Bilirubin (total): Grade 1 | 1 | 0 | 2 | 0 | 0 | 0
  Bilirubin (total): Grade 2 | 1 | 0 | 3 | 1 | 7 | 0
  Bilirubin (total): Grade 3 | 0 | 0 | 2 | 5 | 8 | 10
  Bilirubin (total): Grade 4 | 0 | 0 | 2 | 3 | 1 | 6
  Creatinine (CR): Grade 1 | 9 | 11 | 8 | 6 | 6 | 10
  CR: Grade 2 | 2 | 4 | 7 | 3 | 8 | 5
  CR: Grade 3 | 0 | 0 | 1 | 0 | 1 | 1
  Hyperglycemia: Grade 1 | 5 | 8 | 10 | 8 | 5 | 8
  Hyperglycemia: Grade 2 | 1 | 2 | 5 | 0 | 4 | 2
  Hyperglycemia: Grade 3 | 0 | 1 | 1 | 0 | 0 | 4
  Hyperkalemia: Grade 1 | 2 | 1 | 4 | 2 | 3 | 1
  Hyperkalemia: Grade 2 | 0 | 0 | 1 | 0 | 0 | 0
  Hyperkalemia: Grade 3 | 0 | 0 | 1 | 0 | 1 | 0
  Hypermagnesemia: Grade 1 | 1 | 1 | 4 | 0 | 2 | 3
  Hypoalbuminemia: Grade 1 | 5 | 4 | 2 | 1 | 0 | 0
  Hypoalbuminemia: Grade 2 | 5 | 10 | 9 | 8 | 14 | 8
  Hypoalbuminemia: Grade 3 | 0 | 0 | 3 | 1 | 2 | 7
  Hypocalcemia: Grade 1 | 5 | 11 | 5 | 3 | 4 | 7
  Hypocalcemia: Grade 2 | 3 | 1 | 9 | 4 | 9 | 9
  Hypoglycemia: Grade 1 | 0 | 0 | 2 | 0 | 2 | 2
  Hypokalemia: Grade 1 | 4 | 1 | 5 | 0 | 5 | 4
  Hypokalemia: Grade 3 | 0 | 0 | 0 | 1 | 0 | 0
  Hypomagnesemia: Grade 1 | 0 | 2 | 5 | 3 | 4 | 6
  Hyponatremia: Grade 1 | 5 | 5 | 4 | 5 | 7 | 8
  Hyponatremia: Grade 3 | 1 | 4 | 7 | 5 | 7 | 7
  Hypophosphatemia: Grade 1 | 0 | 3 | 1 | 0 | 0 | 1
  Hypophosphatemia: Grade 2 | 1 | 2 | 3 | 3 | 3 | 3
  Hypophosphatemia: Grade 3 | 2 | 0 | 1 | 1 | 3 | 1

37. Other Pre Specified Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Criteria for abnormal value of ECG parameters: maximum increase from baseline (IFB) in QT interval using Fridericia's correction (QTcF)/QT interval using Bazett's correction (QTcB) range from less than (<)30 millisecond (msec), 30 to <60, greater than or equal to (>=)60 msec; maximum post-dose QTcF/QTcB ranges from <450 msec, 450 to <480 msec, 480 to <500, and >=500 msec; PR interval: >=50 percent (%) increase when baseline <200 msec; or increase >=25% when baseline less than or equal to (<=)200 msec; QRS interval: >=50% increase when baseline <100 msec; >=25% increase when baseline >=100 msec. Only categories which included atleast 1 participant with abnormality are reported in this outcome measure.
Time Frame: Baseline up to end of treatment (up to 728 days)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 11 | 15 | 20 | 10 | 16 | 16
participants
  Maximum Post-dose QTCF Interval: <450 msec | 9 | 13 | 13 | 8 | 11 | 6
  Maximum Post-dose QTCF Interval: 450 to <480 msec | 1 | 2 | 6 | 1 | 5 | 9
  Maximum Post-dose QTCF Interval: 480 to <500 msec | 1 | 0 | 0 | 1 | 0 | 1
  Maximum Post-dose QTCF Interval: >=500 msec | 0 | 0 | 1 | 0 | 0 | 0
  Maximum Post-dose QTCB Interval: <450 msec | 10 | 13 | 12 | 7 | 11 | 5
  Maximum Post-dose QTCB Interval: 450 to <480 msec | 0 | 2 | 7 | 2 | 5 | 8
  Maximum Post-dose QTCB Interval: 480 to <500 msec | 1 | 0 | 0 | 1 | 0 | 1
  Maximum Post-dose QTCB Interval: >=500 msec | 0 | 0 | 1 | 0 | 0 | 2
  Maximum QTCF Interval IFB: <30 msec | 7 | 12 | 11 | 7 | 7 | 8
  Maximum QTCF Interval IFB: 30 to 60 msec | 2 | 1 | 1 | 0 | 4 | 1
  Maximum QTCF IFB: >=60 msec | 0 | 0 | 0 | 1 | 0 | 1
  Maximum QTCB Interval IFB: <30 msec | 7 | 10 | 8 | 5 | 7 | 7
  Maximum QTCB Interval IFB: 30 to 60 msec | 0 | 1 | 0 | 1 | 1 | 1
  Maximum QTCB Interval IFB: >=60 msec | 0 | 0 | 0 | 1 | 0 | 1
  Maximum PR Interval IFB: >=50% | 0 | 1 | 0 | 0 | 0 | 0
  Maximum PR Interval IFB, Other Than: >=25 or 50% | 10 | 14 | 19 | 10 | 15 | 16
  Maximum QRS Interval IFB, Other Than: >=25 or 50% | 11 | 15 | 20 | 10 | 16 | 16

38. Other Pre Specified Outcome: Number of Participants With Abnormal Fundoscopy Examination Findings
Description: Fundoscopy examination included an examination of the vitreous body, retina macula, retina non-macula, optic nerve head, optic disc notching and fundus using the category of the examination status (normal, mild, moderate, or severe). In this outcome measure, number of participants with abnormal fundoscopy values identified by investigator were reported.
Time Frame: Baseline up to end of treatment (up to 728 days)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 11 | 15 | 20 | 10 | 16 | 16
participants
  Right Eye, Retina Macula: Mild Abnormality | 0 | 0 | 1 | 0 | 0 | 0
  Right Eye, Retina Non-Macula: Mild Abnormality | 1 | 0 | 0 | 0 | 0 | 0
  Right Eye, Optic Disc Notching: Mild Abnormality | 1 | 1 | 0 | 0 | 0 | 0
  Right Eye, Fundus: Mild Abnormality | 0 | 0 | 1 | 0 | 0 | 0
  Right Eye, Vitreous Body: Mild Abnormality | 0 | 0 | 0 | 1 | 0 | 0
  Left Eye, Retina Non-Macula: Mild Abnormality | 1 | 0 | 0 | 0 | 1 | 0
  Left Eye, Vitreous Body: Mild Abnormality | 1 | 0 | 0 | 1 | 0 | 0
  Left Eye, Fundus: Mild Abnormality | 0 | 0 | 1 | 0 | 0 | 0
  Left Eye, Retina Macula: Mild Abnormality | 0 | 0 | 1 | 0 | 0 | 0
  Left Eye, Optic Disc Notching: Mild Abnormality | 1 | 0 | 0 | 0 | 0 | 0

39. Other Pre Specified Outcome: Objective Response Rate (ORR)
Description: ORR was defined as percentage of participants with confirmed complete response (CR) or partial response (PR) according to response evaluation criteria in solid tumors (RECIST) version 1.1. In case of target lesions CR was defined as the disappearance of all target lesions and in case nodal disease included in the sum of target lesions. The nodes decreased to normal size (<10 mm). In case of non-target lesions disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Confirmed responses were those who persisted on repeat imaging study at least 4 weeks after the initial documentation of response.
Time Frame: Baseline, every 8 weeks until disease progression or unacceptable toxicity up to end of treatment (up to 728 days)
Population: Response-evaluable population was defined as all participants in the safety analysis population who had an adequate baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 11 | 15 | 20 | 10 | 16 | 16
percentage of participants | 9.1 [0.2 to 41.3] | 0 [0.0 to 21.8] | 5.0 [0.1 to 24.9] | 0 [0.0 to 30.8] | 6.3 [0.2 to 30.2] | 0 [0.0 to 20.6]

40. Other Pre Specified Outcome: Duration of Response (DR)
Description: DR was defined as the time from date of first documentation of CR or PR to first documentation of objective tumor progression or death due to any cause, whichever occurred first. In case of target lesions CR was defined as the disappearance of all target lesions and in case nodal disease included in the sum of target lesions. The nodes decreased to normal size (<10 mm). In case of non-target lesions disappearance of all non-target lesions and normalization of tumor marker level. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Objective tumor progression as per RECIST version 1.1 was defined as >=20% increase in sum of diameters of target lesions taking as a reference smallest sum of diameters recorded since treatment started, or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. DR was estimated using Kaplan-Meier method.
Time Frame: Baseline, every 8 weeks until disease progression or unacceptable toxicity up to end of treatment (up to 728 days)
Population: Response evaluable population. Here, 'N' signifies participants who were evaluable for this outcome measure. Data for normal hepatic function (200 mg), moderate (250 mg) and severe (250 mg) hepatic impairment arms was not estimable since no participants had achieved CR or PR in these reporting arms.
Measure: Median (95% Confidence Interval); unit: week
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
Number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0
week | NA [NA to NA] — Median and 95% CI were not estimable since there were no participant who had event ( disease progression or death) in this reporting group. |  | 17.4 [NA to NA] — 95% CI were not estimable since only 1 participant was evaluable in this reporting group. |  | NA [NA to NA] — Median and 95% CI were not estimable since there were no participant who had event ( disease progression or death) in this reporting group. |

ADVERSE EVENTS:
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Normal Hepatic Function: Crizotinib 250 mg Twice Daily | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily | Severe Hepatic Impairment Crizotinib 250 mg Once Daily
All-Cause Mortality (participants affected / at risk) | 3/11 | 4/15 | 8/20 | 5/10 | 7/16 | 9/16
Serious Adverse Events (participants affected / at risk) | 7/11 | 8/15 | 13/20 | 6/10 | 14/16 | 14/16
Other Adverse Events (participants affected / at risk) | 11/11 | 15/15 | 20/20 | 9/10 | 16/16 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Hepatic Function: Crizotinib 250 mg Twice Daily (N=11) | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily (N=15) | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily (N=20) | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily (N=10) | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily (N=16) | Severe Hepatic Impairment Crizotinib 250 mg Once Daily (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 2 | 2 | 4 | 5 | 4 | 6
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 2
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 2 | 2 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Wound drainage (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Normal Hepatic Function: Crizotinib 250 mg Twice Daily (N=11) | Normal Hepatic Function: Crizotinib 200/250 mg Twice Daily (N=15) | Mild Hepatic Impairment: Crizotinib 250 mg Twice Daily (N=20) | Moderate Hepatic Impairment Crizotinib 200 mg Twice Daily (N=10) | Moderate Hepatic Impairment: Crizotinib 250 mg Once Daily (N=16) | Severe Hepatic Impairment Crizotinib 250 mg Once Daily (N=16)
Anaemia (Blood and lymphatic system disorders) | 3 | 5 | 6 | 2 | 5 | 3
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 2 | 0 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Halo vision (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 2 | 1 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 4 | 1 | 2 | 3 | 2 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 2 | 0 | 2 | 3 | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 0 | 2 | 1 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 5 | 2 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 6 | 2 | 4 | 1 | 4 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 5 | 1 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 8 | 11 | 2 | 7 | 6
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 8 | 6 | 2 | 9 | 3
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 4 | 6 | 4 | 5 | 8 | 7
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 3 | 0
Pain (General disorders) | 1 | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 3 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 4 | 2 | 8 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 3 | 1 | 1 | 1
Oedema peripheral (General disorders) | 4 | 2 | 3 | 3 | 5 | 3
Fall (Injury, poisoning and procedural complications) | 3 | 3 | 1 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 1 | 6 | 1 | 2 | 4
Ammonia increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 4 | 7 | 2 | 5 | 5
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 2 | 2 | 1 | 2 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 5 | 1 | 1
Blood creatinine increased (Investigations) | 5 | 4 | 5 | 4 | 3 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Heart rate decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 3
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1 | 1 | 3
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1 | 2 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 3
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4 | 5 | 2 | 6 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0 | 3 | 2
Food intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 2 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 6 | 5 | 6 | 4 | 6
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 4 | 2 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 1 | 4 | 2
Dysgeusia (Nervous system disorders) | 3 | 2 | 4 | 2 | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 1 | 1 | 1 | 0 | 3
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1
Visual perseveration (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 2 | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 3 | 1 | 0 | 1
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0/7 | 0/9 | 0/13 | 1/8 | 1/10 | 0/10 — This AE was gender specific.
Gynaecomastia (Reproductive system and breast disorders) | 0/7 | 0/9 | 0/13 | 1/8 | 0/10 | 0/10 — This AE was gender specific.
Ovarian cyst (Reproductive system and breast disorders) | 1/4 | 0/6 | 0/7 | 0/2 | 0/6 | 0/6 — This AE was gender specific.
Penile swelling (Reproductive system and breast disorders) | 0/7 | 0/9 | 0/13 | 1/8 | 0/10 | 0/10 — This AE was gender specific.
Scrotal oedema (Reproductive system and breast disorders) | 1/7 | 0/9 | 0/13 | 0/8 | 0/10 | 0/10 — This AE was gender specific.
Scrotal pain (Reproductive system and breast disorders) | 1/7 | 0/9 | 0/13 | 0/8 | 0/10 | 0/10 — This AE was gender specific.
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/4 | 0/6 | 0/7 | 0/2 | 0/6 | 1/6 — This AE was gender specific.
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1 | 1 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 2 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 3 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.